CLINICAL TRIAL: NCT06677840
Title: Precision Health in Autism: Exploring the Gut-Brain-Behavior Axis With Biomarkers, Probiotic Efficacy, and Artificial Intelligence Algorithms
Brief Title: Exploring the Gut-Brain-Behavior Axis With Biomarkers, Probiotic Efficacy, and Artificial Intelligence Algorithms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202404049RIPA
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GKB7 (Experimental)
  Interventions: Other: probiotic (GKB7/placebo)
- Placebo (Placebo Comparator)
  Interventions: Other: probiotic (GKB7/placebo)

INTERVENTIONS:
Other: probiotic (GKB7/placebo) — The objectives of this double-blind randomized placebo-controlled trial are to evaluate the tolerability, safety, and efficacy of the probiotic intervention with Clostridium butyricum GKB7 among 90 4-15-year-old children and adolescents with a clinical diagnosis of ASD according to the DSM-5

SUMMARY:
This groundbreaking human study on the ASD microbiome includes probiotic clinical trials, investigation of treatment biomarkers, machine learning/deep learning platform development for ASD classification and prediction, and identification of diagnostic biomarkers. Upon completion, the investigators anticipate publishing at least 12 SCI papers and/or patents and establishing an auxiliary diagnosis platform for both clinical and academic purposes. The findings will offer new insights into the pathogenetic mechanisms, improving early detection, diagnosis, and treatment, ultimately advancing precision medicine for ASD.

DETAILED DESCRIPTION:
With an increased prevalence of autism spectrum disorder (ASD) worldwide and in Taiwan, ASD demands urgent attention due to its lasting impact, unclear causes, and limited diagnostic and treatment options. Recent studies highlight disruptions in the gut-brain axis, particularly in ASD. Building on PI Gau's prior research on altered gut microbiota in autism spectrum disorder (ASD), this proposed 4-year study aims to develop evidence-based probiotic intervention (GKB7) and treatment biomarkers for behavioral interventions (Naturalistic Developmental Behavioral Interventions, NDBI, and Program for the Education and Enrichment of Relational Skills, PEERS®) through comprehensive assessments. The ultimate goal is to establish probiotic treatments and diagnostic/treatment biomarkers for ASD utilizing a deep-learning multimodal auxiliary platform.

Specific Aims:

S.I To conduct a randomized, double-blind, placebo-controlled trial to assess the treatment effects of Clostridium butyricum GKB7 on ASD.

S.II To investigate the effect of NDBI intervention trials using metagenomics as the outcome measure.

S.III To evaluate the effect of PEERS® interventional trials with metagenomics as the outcome measure.

S.IV To develop an artificial intelligence (machine/deep learning) multimodal auxiliary prediction platform that integrates environmental, behavioral/clinical, neurocognitive/imaging, and metagenomic data for ASD diagnosis, subtyping, and impairment prediction.

S.V To identify microbiome and metabolomic biomarkers and endophenotypes of ASD, and to establish Gut-Brain-Behavioral Axes in ASD.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 4 to 15 who are clinically diagnosed with ASD according to DSM-5 criteria and confirmed by the ADI-R/ADOS.
* Caregivers cooperate with all the assessments and stool and blood collection.

Exclusion Criteria:

* A history of major psychiatric disorders (e.g., schizophrenia, bipolar disorder, major depression), neurological disorders, and substances use disorders.
* Difficulty following instructions.
* Consumption of antibiotics and yogurt or probiotic products two weeks prior to enrollment.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression | At baseline (before treatment, V0), month 1 (V1), month 2 (V2), month 3 (V3), month 4 (V4), and month 6 (V5)
  The CGI-S (Clinical Global Impression-Severity Scale) and CGI-I (-Improvement Scale) are single-item ratings of the clinician's assessment of the global severity of clinical symptoms. Severity and improvement are rated on a 7-point scale (from 1 = normal, not at all ill, to 7 = among the most extremely ill) and (from 1 = very much improved, to 7 = very much worse).
Social Responsiveness Scale (SRS) | At baseline (before treatment, V0), month 1 (V1), month 2 (V2), month 3 (V3), month 4 (V4), and month 6 (V5)
  The SRS is a 65-item questionnaire based on parent-reports on the child's social interactions with others (rating 0-3), consists of 5 subscales: social awareness, social cognition, social communication, social motivation, and autistic mannerisms

SECONDARY OUTCOMES:
Self-administered questionnaires | At baseline (before treatment, V0), month 3 (V3), and month 6 (V5)
  The self-administered questionnaires include autistic symptoms (Autism Spectrum Quotient, AQ; Sensory Profile, SP), psychopathology (Child Behavior Checklist, CBCL; Swanson, Nolan, and Pelham, version IV scale, SNAP-IV), social functions/quality of life (Social Adjustment Inventory for Children and Adolescents, SAICA), and executive functions (Behavior Rating Inventories of Executive Function, BRIEF)
Neuropsychological functions: Continuous Performance Test(CPT) | At baseline (before treatment, V0), month 3 (V3), and month 6 (V5)
  The 4 dimensions of CCPT: focused attention, hyperactivity/impulsivity, sustained attention, and vigilance
Neuropsychological functions: Cambridge Neuropsychological Test Automated Batteries(CANTAB) | At baseline (before treatment, V0), month 3 (V3), and month 6 (V5)
  The 4 main cognitive components of CANTAB: Visual Memory, Attention, Working and Planning Memory (Executive Functions), and Decision Making

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan